CLINICAL TRIAL: NCT01159600
Title: A Phase III Randomised, Double-blind, Placebo-controlled, Parallel Group, Efficacy and Safety Study of BI 10773 (10 mg, 25 mg) Administered Orally, Once Daily Over 24 Weeks in Patients With Type 2 Diabetes Mellitus With Insufficient Glycaemic Control Despite Treatment With Metformin Alone or Metformin in Combination With a Sulfonylurea
Brief Title: Efficacy and Safety Study With Empagliflozin (BI 10773) vs. Placebo as add-on to Metformin or Metformin Plus Sulfonylurea Over 24 Weeks in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.23; 2009-016258-41 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (4):
- BI 10773 Arm 2 (Experimental): BI 10773 once daily high dose
  Interventions: Drug: BI 10773; Drug: Placebo identical to BI 10773 low dose
- Placebo (Placebo Comparator): Placebo matching BI 10773
  Interventions: Drug: Placebo identical to BI 10773 low dose; Drug: Placebo identical to BI 10773 high dose
- BI 10773 open-label (Experimental): BI 10773 once daily high dose open label
  Interventions: Drug: BI 10773
- BI 10773 Arm 1 (Experimental): BI 10773 once daily low dose
  Interventions: Drug: Placebo identical to BI 10773 high dose; Drug: BI 10773

INTERVENTIONS:
Drug: Placebo identical to BI 10773 high dose — Placebo tablets matching BI 10773 high dose
  Arms: BI 10773 Arm 1
Drug: Placebo identical to BI 10773 low dose — Placebo tablets matching BI 10773 low dose
  Arms: Placebo
Drug: BI 10773 — BI 10773 tablets once daily high dose open label
  Arms: BI 10773 open-label
Drug: BI 10773 — BI 10773 tablets once daily high dose
  Arms: BI 10773 Arm 2
Drug: Placebo identical to BI 10773 low dose — Placebo tablets matching BI 10773 low dose
  Arms: BI 10773 Arm 2
Drug: BI 10773 — BI 10773 tablets once daily low dose
  Arms: BI 10773 Arm 1
Drug: Placebo identical to BI 10773 high dose — Placebo tablets matching BI 10773 high dose
  Arms: Placebo

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of two doses of BI 10773 compared to placebo given for 24 weeks as add-on therapy to metformin or metformin plus sulfonylurea in patients with Typ 2 Diabetes Mellitus with insufficient glycaemic control.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of type 2 diabetes mellitus prior to informed consent
2. Male and female patients on a diet and exercise regimen who are pre-treated with immediate release metformin or immediate release metformin plus sulfonylurea (see below for minimum doses). The treatment regimen has to be unchanged for 12 weeks prior to randomisation.

   Minimum dose for metformin: > or = 1500 mg/day or maximum tolerated dose or maximum dose according to local label Minimum dose for sulfonylurea: > or = half of the maximal recommended dose or maximum tolerated dose or maximum dose according to local label
3. HbA1c of > or = 7.0% and < or = 11% at Visit 1 (screening) in order to be eligible for randomised treatment HbA1c of > 11% at Visit 1 (screening) in order to be eligible for the open-label treatment arm (25 mg BI 10773)
4. Age> or = 18
5. Body Mass Index (BM)I < or = 45 kg/m2 (Body Mass Index) at Visit 1 (Screening)
6. Signed and dated written informed consent by date of Visit 1 in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

1. Uncontrolled hyperglycaemia with a glucose level > 240 mg/dl (>13.3 mmol/L) after an overnight fast during placebo run-in and confirmed by a second measurement (not on the same day)
2. Any other antidiabetic drug within 12 weeks prior to randomisation except those mentioned in inclusion criterion 2
3. Myocardial infarction, stroke or transient ischemic attack (TIA) within 3 months prior to informed consent
4. Indication of liver disease, defined by serum levels of either ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined during screening and/or run-in phase
5. Impaired renal function, defined as eGFR<30 ml/min (severe renal impairment) as determined during screening and/or run-in phase
6. Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption
7. Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years
8. Contraindications to metformin and/or sulfonylurea according to the local label for those patients that enter the study with the respective background therapy
9. Blood dyscrasias or any disorders causing haemolysis or unstable Red Blood Cell (e.g. malaria, babesiosis, haemolytic anaemia)
10. Treatment with anti-obesity drugs (e.g. sibutramine, orlistat) 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight
11. Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except Typ 2 Diabetes
12. Pre-menopausal women (last menstruation ¿ 1 year prior to informed consent) who:

    * are nursing or pregnant or
    * are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence (if acceptable by local authorities), double barrier method and vasectomised partner
13. Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake
14. Participation in another trial with an investigational drug within 30 days prior to informed consent
15. Any other clinical condition that would jeopardize patients safety while participating in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1504 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (148):
- United States (25):
  - 1245.23.10145 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1245.23.10046 Boehringer Ingelheim Investigational Site, Tempe, Arizona
  - 1245.23.10095 Boehringer Ingelheim Investigational Site, Huntington Park, California
  - 1245.23.10109 Boehringer Ingelheim Investigational Site, Huntington Park, California
  - 1245.23.10074 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1245.23.10149 Boehringer Ingelheim Investigational Site, Rancho Cucamonga, California
  - 1245.23.10127 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1245.23.10042 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1245.23.10133 Boehringer Ingelheim Investigational Site, Jupiter, Florida
  - 1245.23.10080 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1245.23.10001 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1245.23.10159 Boehringer Ingelheim Investigational Site, Des Moines, Iowa
  - 1245.23.10117 Boehringer Ingelheim Investigational Site, Arkansas City, Kansas
  - 1245.23.10157 Boehringer Ingelheim Investigational Site, Newton, Kansas
  - 1245.23.10148 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 1245.23.10034 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1245.23.10123 Boehringer Ingelheim Investigational Site, Smithtown, New York
  - 1245.23.10120 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1245.23.10031 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1245.23.10158 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 1245.23.10015 Boehringer Ingelheim Investigational Site, Simpsonville, South Carolina
  - 1245.23.10156 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.23.10153 Boehringer Ingelheim Investigational Site, Hurst, Texas
  - 1245.23.10143 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1245.23.10106 Boehringer Ingelheim Investigational Site, San Antonio, Texas
- Canada (21):
  - 1245.23.20032 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1245.23.20023 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1245.23.20028 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1245.23.20033 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1245.23.20024 Boehringer Ingelheim Investigational Site, Paradise, Newfoundland and Labrador
  - 1245.23.20031 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1245.23.20026 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1245.23.20001 Boehringer Ingelheim Investigational Site, Barrie, Ontario
  - 1245.23.20022 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1245.23.20035 Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - 1245.23.20030 Boehringer Ingelheim Investigational Site, Etobicoke, Ontario
  - 1245.23.20037 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1245.23.20029 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1245.23.20003 Boehringer Ingelheim Investigational Site, Markham, Ontario
  - 1245.23.20040 Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - 1245.23.20034 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1245.23.20039 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1245.23.20027 Boehringer Ingelheim Investigational Site, Laval, Quebec
  - 1245.23.20025 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1245.23.20038 Boehringer Ingelheim Investigational Site, Saint-Laurent, Quebec
  - 1245.23.20036 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
- China (26):
  - 1245.23.86031 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.23.86032 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.23.86033 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.23.86034 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.23.86035 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.23.86048 Boehringer Ingelheim Investigational Site, Chengdu
  - 1245.23.86058 Boehringer Ingelheim Investigational Site, Chongqing
  - 1245.23.86038 Boehringer Ingelheim Investigational Site, Dalian
  - 1245.23.86002 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1245.23.86052 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1245.23.86037 Boehringer Ingelheim Investigational Site, Haerbin
  - 1245.23.86049 Boehringer Ingelheim Investigational Site, Jinan
  - 1245.23.86053 Boehringer Ingelheim Investigational Site, Jinan
  - 1245.23.86042 Boehringer Ingelheim Investigational Site, Nanjing
  - 1245.23.86043 Boehringer Ingelheim Investigational Site, Nanjing
  - 1245.23.86055 Boehringer Ingelheim Investigational Site, Nanning
  - 1245.23.86056 Boehringer Ingelheim Investigational Site, Nanning
  - 1245.23.86039 Boehringer Ingelheim Investigational Site, Shanghai
  - 1245.23.86040 Boehringer Ingelheim Investigational Site, Shanghai
  - 1245.23.86054 Boehringer Ingelheim Investigational Site, Shantou
  - 1245.23.86057 Boehringer Ingelheim Investigational Site, Shenyang
  - 1245.23.86045 Boehringer Ingelheim Investigational Site, Shijiazhuang
  - 1245.23.86013 Boehringer Ingelheim Investigational Site, Suzhou
  - 1245.23.86036 Boehringer Ingelheim Investigational Site, Tianjin
  - 1245.23.86041 Boehringer Ingelheim Investigational Site, Xi'an
  - 1245.23.86051 Boehringer Ingelheim Investigational Site, Zhenjiang
- France (17):
  - 1245.23.33015 Boehringer Ingelheim Investigational Site, Arras
  - 1245.23.33008 Boehringer Ingelheim Investigational Site, Bersée
  - 1245.23.33020 Boehringer Ingelheim Investigational Site, Bischheim
  - 1245.23.33002 Boehringer Ingelheim Investigational Site, Bondy
  - 1245.23.33016 Boehringer Ingelheim Investigational Site, Bruay-la-Buissière
  - 1245.23.33001 Boehringer Ingelheim Investigational Site, Corbeil-Essonnes
  - 1245.23.33010 Boehringer Ingelheim Investigational Site, Croix
  - 1245.23.33009 Boehringer Ingelheim Investigational Site, Hautmont
  - 1245.23.33003 Boehringer Ingelheim Investigational Site, La Rochelle
  - 1245.23.33045 Boehringer Ingelheim Investigational Site, Marseille
  - 1245.23.33014 Boehringer Ingelheim Investigational Site, Mundolsheim
  - 1245.23.33004 Boehringer Ingelheim Investigational Site, Narbonne
  - 1245.23.33012 Boehringer Ingelheim Investigational Site, Schiltigheim
  - 1245.23.33013 Boehringer Ingelheim Investigational Site, Strasbourg
  - 1245.23.33019 Boehringer Ingelheim Investigational Site, Strasbourg
  - 1245.23.33007 Boehringer Ingelheim Investigational Site, Vieux-Condé
  - 1245.23.33018 Boehringer Ingelheim Investigational Site, Wattrelos
- Germany (11):
  - 1245.23.49001 Boehringer Ingelheim Investigational Site, Dormagen
  - 1245.23.49009 Boehringer Ingelheim Investigational Site, Flörsheim
  - 1245.23.49004 Boehringer Ingelheim Investigational Site, Hatten
  - 1245.23.49007 Boehringer Ingelheim Investigational Site, Künzing
  - 1245.23.49002 Boehringer Ingelheim Investigational Site, Neuwied
  - 1245.23.49008 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1245.23.49010 Boehringer Ingelheim Investigational Site, Rednitzhembach
  - 1245.23.49006 Boehringer Ingelheim Investigational Site, Rehburg-Loccum
  - 1245.23.49011 Boehringer Ingelheim Investigational Site, Rehlingen-Siersburg
  - 1245.23.49005 Boehringer Ingelheim Investigational Site, Saarbrücken
  - 1245.23.49003 Boehringer Ingelheim Investigational Site, Unterschneidheim
- India (5):
  - 1245.23.91101 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1245.23.91104 Boehringer Ingelheim Investigational Site, Indore
  - 1245.23.91103 Boehringer Ingelheim Investigational Site, Maharashtra
  - 1245.23.91102 Boehringer Ingelheim Investigational Site, Nagpur
  - 1245.23.91105 Boehringer Ingelheim Investigational Site, Pune
- Mexico (4):
  - 1245.23.52003 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1245.23.52004 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1245.23.52001 Boehringer Ingelheim Investigational Site, Monterrey
  - 1245.23.52002 Boehringer Ingelheim Investigational Site, Monterrey
- Slovakia (7):
  - 1245.23.74005 Boehringer Ingelheim Investigational Site, Bratislava
  - 1245.23.74002 Boehringer Ingelheim Investigational Site, Lučenec
  - 1245.23.74006 Boehringer Ingelheim Investigational Site, Nitra
  - 1245.23.74014 Boehringer Ingelheim Investigational Site, Nové Zámky
  - 1245.23.74001 Boehringer Ingelheim Investigational Site, Považská Bystrica
  - 1245.23.74004 Boehringer Ingelheim Investigational Site, Prešov
  - 1245.23.74003 Boehringer Ingelheim Investigational Site, Trebišov
- Slovenia (3):
  - 1245.23.38003 Boehringer Ingelheim Investigational Site, Celje
  - 1245.23.38002 Boehringer Ingelheim Investigational Site, Koper
  - 1245.23.38001 Boehringer Ingelheim Investigational Site, Maribor
- South Korea (13):
  - 1245.23.82012 Boehringer Ingelheim Investigational Site, Anyang
  - 1245.23.82004 Boehringer Ingelheim Investigational Site, Busan
  - 1245.23.82011 Boehringer Ingelheim Investigational Site, Goyang
  - 1245.23.82009 Boehringer Ingelheim Investigational Site, Ilsan
  - 1245.23.82001 Boehringer Ingelheim Investigational Site, Incheon
  - 1245.23.82006 Boehringer Ingelheim Investigational Site, Jeonju
  - 1245.23.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.23.82007 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.23.82008 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.23.82010 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.23.82014 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.23.82002 Boehringer Ingelheim Investigational Site, Suwon
  - 1245.23.82003 Boehringer Ingelheim Investigational Site, Wŏnju
- Taiwan (10):
  - 1245.23.88010 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.23.88011 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.23.88012 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.23.88013 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.23.88009 Boehringer Ingelheim Investigational Site, Taichung
  - 1245.23.88014 Boehringer Ingelheim Investigational Site, Tainan
  - 1245.23.88006 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.23.88007 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.23.88021 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.23.88008 Boehringer Ingelheim Investigational Site, Taoyuan
- Turkey (Türkiye) (6):
  - 1245.23.90003 Boehringer Ingelheim Investigational Site, Erzurum
  - 1245.23.90001 Boehringer Ingelheim Investigational Site, Gaziantep
  - 1245.23.90002 Boehringer Ingelheim Investigational Site, Istanbul
  - 1245.23.90006 Boehringer Ingelheim Investigational Site, Istanbul
  - 1245.23.90007 Boehringer Ingelheim Investigational Site, Istanbul
  - 1245.23.90004 Boehringer Ingelheim Investigational Site, Izmir

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Inzucchi SE, Davies MJ, Khunti K, Trivedi P, George JT, Zwiener I, Johansen OE, Sattar N. Empagliflozin treatment effects across categories of baseline HbA1c, body weight and blood pressure as an add-on to metformin in patients with type 2 diabetes. Diabetes Obes Metab. 2021 Feb;23(2):425-433. doi: 10.1111/dom.14234. Epub 2020 Nov 20. PMID 33084149
- [Derived] Cherney D, Lund SS, Perkins BA, Groop PH, Cooper ME, Kaspers S, Pfarr E, Woerle HJ, von Eynatten M. The effect of sodium glucose cotransporter 2 inhibition with empagliflozin on microalbuminuria and macroalbuminuria in patients with type 2 diabetes. Diabetologia. 2016 Sep;59(9):1860-70. doi: 10.1007/s00125-016-4008-2. Epub 2016 Jun 17. PMID 27316632
- [Derived] Haring HU, Merker L, Seewaldt-Becker E, Weimer M, Meinicke T, Woerle HJ, Broedl UC; EMPA-REG METSU Trial Investigators. Empagliflozin as add-on to metformin plus sulfonylurea in patients with type 2 diabetes: a 24-week, randomized, double-blind, placebo-controlled trial. Diabetes Care. 2013 Nov;36(11):3396-404. doi: 10.2337/dc12-2673. Epub 2013 Aug 20. PMID 23963895

RESULTS

PARTICIPANT FLOW:
Groups:
- Met: Placebo: A placebo tablet, matching the empagliflozin 10mg and 25mg tablets, taken once daily for 24 weeks in patients with background medication of metformin only.
- Met: Empa 10mg: Single oral dose of empagliflozin (empa) 10mg taken once daily for 24 weeks in patients with background medication of metformin only.
- Met: Empa 25mg; Met: Empa 25mg Open Label: Single oral dose of empagliflozin (empa) 25mg taken once daily for 24 weeks in patients with background medication of metformin only.
- Met+SU: Placebo: A placebo tablet, matching the empagliflozin 10mg and 25mg tablets, taken once daily for 24 weeks in patients with background medication of metformin plus sulphonylurea (SU).
- Met+SU: Empa 10mg: Single oral dose of empagliflozin (empa) 10mg taken once daily for 24 weeks in patients with background medication of metformin plus sulphonylurea (SU).
- Met+SU: Empa 25mg; Met+SU: Empa 25mg Open Label: Single oral dose of empagliflozin (empa) 25mg taken once daily for 24 weeks in patients with background medication of metformin plus sulphonylurea (SU).
Period: Overall Study
Arm/Group | Met: Placebo | Met: Empa 10mg | Met: Empa 25mg | Met: Empa 25mg Open Label | Met+SU: Placebo | Met+SU: Empa 10mg | Met+SU: Empa 25mg | Met+SU: Empa 25mg Open Label
Started | 207 | 217 | 214 | 69 | 225 | 226 | 218 | 103
Completed | 186 | 209 | 196 | 58 | 201 | 208 | 199 | 85
Not Completed | 21 | 8 | 18 | 11 | 24 | 18 | 19 | 18
Not completed — Not treated | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2
Not completed — Adverse Event | 7 | 2 | 5 | 1 | 8 | 6 | 7 | 5
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Non compliant with protocol | 2 | 1 | 0 | 0 | 2 | 0 | 2 | 0
Not completed — Lost to Follow-up | 2 | 3 | 4 | 3 | 3 | 0 | 3 | 2
Not completed — Patient refusal to continue,not due toAE | 7 | 2 | 4 | 5 | 4 | 4 | 2 | 5
Not completed — Other reason not defined above | 3 | 0 | 4 | 2 | 5 | 7 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS), which included all randomised patients treated with at least one dose of study drug with a baseline HbA1c value. Treatment assignment as randomised.
  Open label set which included all patients entered in the empa 25mg open-label arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Met: Placebo | Met: Empa 10mg | Met: Empa 25mg | Met: Empa 25mg Open Label | Met+SU: Placebo | Met+SU: Empa 10mg | Met+SU: Empa 25mg | Met+SU: Empa 25mg Open Label | Total
Number analyzed (Participants) | 207 | 217 | 213 | 69 | 225 | 225 | 216 | 101 | 1473
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (9.7) | 55.5 (9.9) | 55.6 (10.2) | 49.8 (11.5) | 56.9 (9.2) | 57.0 (9.2) | 57.4 (9.3) | 53.4 (10.5) | 55.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 92 | 93 | 28 | 113 | 112 | 102 | 47 | 678
  Male | 116 | 125 | 120 | 41 | 112 | 113 | 114 | 54 | 795

OUTCOME MEASURES:

1. Secondary Outcome: Body Weight Change From Baseline
Description: Body weight change from baseline after 24 weeks.
  For open-label groups the descriptive mean is provided, for randomised groups adjusted means are provided. The means are adjusted separately for metformin alone and metformin plus sulphonylurea background medication.
Time Frame: Baseline and 24 weeks
Population: Full analysis set. Treatment assignment as randomised.
  Open-label analysis: Open-label set which included all patients entered in the empa 25mg open-label treatment arm.
  Values after start of antidiabetic rescue therapy were set to missing and last observation carried forward (LOCF) was used for imputation of missing values.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Met: Placebo | Met: Empa 10mg | Met: Empa 25mg | Met: Empa 25mg Open Label | Met+SU: Placebo | Met+SU: Empa 10mg | Met+SU: Empa 25mg | Met+SU: Empa 25mg Open Label
Number analyzed (Participants) | 207 | 217 | 213 | 69 | 225 | 225 | 216 | 101
kg | -0.45 (0.17) | -2.08 (0.17) | -2.46 (0.17) | -1.33 (0.43) | -0.39 (0.15) | -2.16 (0.15) | -2.39 (0.16) | -1.29 (0.30)
Statistical Analysis 1: Comparison: Met: Placebo vs Met: Empa 10mg; Null hypothesis: No difference in change from baseline to week 24 in body weight between Empagliflozin 10mg and placebo. A hierarchical testing approach was applied to each of the two dose comparisons (10mg vs placebo and 25mg vs placebo) within each background therapy group (metformin and metformin + SU). If for a specific dose the null hypothesis was rejected for the primary endpoint, the same dose was tested against placebo for the change from baseline in body weight; Test type: Superiority or Other; p < 0.0001, ANCOVA — Each of the hypotheses (10mg vs placebo and 25mg vs placebo) were tested (two-sided test) at the significance level of 0.025; ANCOVA with baseline HbA1c and baseline body weight as linear covariates and baseline eGFR, geographical region and treatment as fixed effects; Mean difference = -1.63, 97.5% CI 2-sided [-2.17 to -1.08], Standard Error of Mean 0.24 — Difference calculated as Met: empa 10mg minus Met: placebo
Statistical Analysis 2: Comparison: Met: Placebo vs Met: Empa 25mg; Null hypothesis: No difference in change from baseline to week 24 in body weight between Empagliflozin 25mg and placebo. A hierarchical testing approach was applied to each of the two dose comparisons (10mg vs placebo and 25mg vs placebo) within each background therapy group (metformin and metformin + SU). If for a specific dose the null hypothesis was rejected for the primary endpoint, the same dose was tested against placebo for the change from baseline in body weight; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean difference = -2.01, 97.5% CI 2-sided [-2.56 to -1.46], Standard Error of Mean 0.24 — Difference calculated as Met: empa 25mg minus Met: placebo
Statistical Analysis 3: Comparison: Met+SU: Placebo vs Met+SU: Empa 10mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean difference = -1.76, 97.5% CI 2-sided [-2.25 to -1.28], Standard Error of Mean 0.22 — Difference calculated as Met+SU: empa 10mg minus Met+SU: placebo
Statistical Analysis 4: Comparison: Met+SU: Placebo vs Met+SU: Empa 25mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean difference = -1.99, 97.5% CI 2-sided [-2.48 to -1.50], Standard Error of Mean 0.22 — Difference calculated as Met+SU: empa 25mg minus Met+SU: placebo

2. Secondary Outcome: Mean Daily Plasma Glucose (MDG) Change From Baseline
Description: Change from baseline in mean daily glucose (MDG) using the 8-point blood glucose profile, after 24 weeks of treatment.
  For open-label groups the descriptive mean is provided, for randomised groups adjusted means are provided. The means are adjusted separately for metformin alone and metformin plus sulphonylurea background medication.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Met: Placebo | Met: Empa 10mg | Met: Empa 25mg | Met: Empa 25mg Open Label | Met+SU: Placebo | Met+SU: Empa 10mg | Met+SU: Empa 25mg | Met+SU: Empa 25mg Open Label
Number analyzed (Participants) | 133 | 148 | 147 | 43 | 151 | 148 | 117 | 52
mg/dL | -1.99 (1.99) | -9.64 (1.89) | -14.36 (1.89) | -35.47 (7.34) | 0.00 (1.78) | -10.01 (1.80) | -13.06 (2.03) | -29.34 (6.58)
Statistical Analysis 1: Comparison: Met: Placebo vs Met: Empa 10mg; Null hypothesis (H0): No difference in change from baseline to week 24 in MDG between Empa 10mg and placebo. A hierarchical testing approach was applied to each of the two dose comparisons within each background therapy group. If for a specific dose H0 was rejected for the primary endpoint, the same dose was tested against placebo for change from baseline in body weight. If superiority over placebo was shown at this gate level, then testing proceeded to change from baseline in MDG with that dose; Test type: Superiority or Other; p = 0.0055, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on ANCOVA with baseline HbA1c and baseline MDG as linear covariates and baseline eGFR, geographical region and treatment as fixed effects; Mean difference = -7.65, 97.5% CI 2-sided [-13.81 to -1.48], Standard Error of Mean 2.74 — Difference calculated as Met: empa 10mg minus Met: placebo
Statistical Analysis 2: Comparison: Met: Placebo vs Met: Empa 25mg; Null hypothesis (H0): No difference in change from baseline to week 24 in MDG between Empa 25mg and placebo. A hierarchical testing approach was applied to each of the two dose comparisons within each background therapy group. If for a specific dose H0 was rejected for the primary endpoint, the same dose was tested against placebo for change from baseline in body weight. If superiority over placebo was shown at this gate level, then testing proceeded to change from baseline in MDG with that dose; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean difference = -12.37, 97.5% CI 2-sided [-18.55 to -6.19], Standard Error of Mean 2.75 — Difference calculated as Met: empa 25mg minus Met: placebo
Statistical Analysis 3: Comparison: Met+SU: Placebo vs Met+SU: Empa 10mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean difference = -10.02, 97.5% CI 2-sided [-15.72 to -4.32], Standard Error of Mean 2.53 — Difference calculated as Met+SU: empa 10mg minus Met+SU: placebo
Statistical Analysis 4: Comparison: Met+SU: Placebo vs Met+SU: Empa 25mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean difference = -13.06, 97.5% CI 2-sided [-19.15 to -6.98], Standard Error of Mean 2.70 — Difference calculated as Met+SU: empa 25mg minus Met+SU: placebo

3. Primary Outcome: HbA1c Change From Baseline
Description: Change from baseline in HbA1c after 24 weeks.
  For open-label groups the descriptive mean is provided, for randomised groups adjusted means are provided. The means are adjusted separately for metformin alone and metformin plus sulphonylurea background medication.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of HbA1c
Groups:
- Met: Placebo: A placebo tablet, matching the empagliflozin 10mg and 25mg tablets, taken once daily for 24 weeks, in patients with background medication of metformin only.
Arm/Group | Met: Placebo | Met: Empa 10mg | Met: Empa 25mg | Met: Empa 25mg Open Label | Met+SU: Placebo | Met+SU: Empa 10mg | Met+SU: Empa 25mg | Met+SU: Empa 25mg Open Label
Number analyzed (Participants) | 207 | 217 | 213 | 69 | 225 | 225 | 216 | 101
percentage of HbA1c | -0.13 (0.05) | -0.70 (0.05) | -0.77 (0.05) | -2.78 (0.21) | -0.17 (0.05) | -0.82 (0.05) | -0.77 (0.05) | -2.53 (0.15)
Statistical Analysis 1: Comparison: Met: Placebo vs Met: Empa 10mg; Null hypothesis: No difference in change from baseline to week 24 in HbA1c between Empagliflozin 10mg and placebo. The study consisted of two substudies as defined by the two background medications 'metformin' and 'metformin + SU'. Within each group of background medication, each of the two hypotheses (10mg vs placebo and 25mg vs. placebo) was tested in a two-sided test; Test type: Superiority or Other; p < 0.0001, ANCOVA — Each of the hypotheses (10mg vs placebo and 25mg vs. placebo) were tested (two-sided test) at the significance level of 0.025; Based on ANCOVA with baseline HbA1c as a linear covariate and baseline eGFR (renal function), geographical region and treatment as fixed effects; Mean difference = -0.57, 97.5% CI 2-sided [-0.72 to -0.42], Standard Error of Mean 0.07 — Difference calculated as Met: empa 10mg minus Met: placebo
Statistical Analysis 2: Comparison: Met: Placebo vs Met: Empa 25mg; Null hypothesis: No difference in change from baseline to week 24 in HbA1c between Empagliflozin 25mg and placebo. The study consisted of two substudies as defined by the two background medications 'metformin' and 'metformin + SU'. Within each group of background medication, each of the two hypotheses (10mg vs placebo and 25mg vs. placebo) was tested in a two-sided test; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Based on ANCOVA with baseline HbA1c as a linear covariate and baseline eGFR, geographical region and treatment as fixed effects; Mean difference = -0.64, 97.5% CI 2-sided [-0.79 to -0.48], Standard Error of Mean 0.07 — Difference calculated as Met: empa 25mg minus Met: placebo
Statistical Analysis 3: Comparison: Met+SU: Placebo vs Met+SU: Empa 10mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 2]; Mean difference = -0.64, 97.5% CI 2-sided [-0.79 to -0.49], Standard Error of Mean 0.07 — Difference calculated as Met+SU: empa 10mg minus Met+SU: placebo
Statistical Analysis 4: Comparison: Met+SU: Placebo vs Met+SU: Empa 25mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 2]; Mean difference = -0.59, 97.5% CI 2-sided [-0.74 to -0.44], Standard Error of Mean 0.07 — Difference calculated as Met+SU: empa 25mg minus Met+SU: placebo

4. Other Pre Specified Outcome: Confirmed Hypoglycaemic Adverse Events
Description: Number of patients with confirmed hypoglycaemic events, as reported as adverse events.
Time Frame: From first intake of randomised trial medication until 7 days after last trial medication intake, up to 231 days
Population: Treated set, which included all patients treated with at least one dose of randomised trial medication. Treatment assignment as first medication taken.
  Open label set which included all patients entered into the open-label arm.
Measure: Number; unit: percentage of participants
Arm/Group | Met: Placebo | Met: Empa 10mg | Met: Empa 25mg | Met: Empa 25mg Open Label | Met+SU: Placebo | Met+SU: Empa 10mg | Met+SU: Empa 25mg | Met+SU: Empa 25mg Open Label
Number analyzed (Participants) | 206 | 217 | 214 | 69 | 225 | 224 | 217 | 101
percentage of participants | 0.5 (0.01) | 1.8 (0.01) | 1.4 (0.03) | 2.9 (0.02) | 8.4 (0.01) | 16.1 (0.01) | 11.5 (0.03) | 6.9 (0.02)

ADVERSE EVENTS:
Time Frame: From first intake of randomised trial medication until 7 days after last trial medication intake, up to 231 days
Description: Treated set which included all patients treated with at least one dose of randomised trial medication. Treatment assignment as first medication taken.
  Open label set which included all patients entered into the open-label arm
Arm/Group | Met: Placebo | Met: Empa 10mg | Met: Empa 25mg | Met: Empa 25mg Open Label | Met+SU: Placebo | Met+SU: Empa 10mg | Met+SU: Empa 25mg | Met+SU: Empa 25mg Open Label
Serious Adverse Events (participants affected / at risk) | 7/206 | 7/217 | 5/214 | 1/69 | 14/225 | 11/224 | 1/217 | 5/101
Other Adverse Events (participants affected / at risk) | 56/206 | 29/217 | 38/214 | 18/69 | 76/225 | 77/224 | 67/217 | 28/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Met: Placebo (N=206) | Met: Empa 10mg (N=217) | Met: Empa 25mg (N=214) | Met: Empa 25mg Open Label (N=69) | Met+SU: Placebo (N=225) | Met+SU: Empa 10mg (N=224) | Met+SU: Empa 25mg (N=217) | Met+SU: Empa 25mg Open Label (N=101)
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Listeria sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syringomyelia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Met: Placebo (N=206) | Met: Empa 10mg (N=217) | Met: Empa 25mg (N=214) | Met: Empa 25mg Open Label (N=69) | Met+SU: Placebo (N=225) | Met+SU: Empa 10mg (N=224) | Met+SU: Empa 25mg (N=217) | Met+SU: Empa 25mg Open Label (N=101)
Nasopharyngitis (Infections and infestations) | 16 | 12 | 15 | 5 | 11 | 18 | 13 | 5
Urinary tract infection (Infections and infestations) | 8 | 9 | 9 | 5 | 15 | 21 | 15 | 3
Upper respiratory tract infections (Infections and infestations) | 9 | 2 | 9 | 4 | 12 | 7 | 11 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 22 | 35 | 28 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 23 | 5 | 2 | 2 | 28 | 6 | 5 | 8
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 3 | 4 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 12 | 5 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.